CLINICAL TRIAL: NCT01683214
Title: Potential Use of Brain Network Activation (BNA) Analysis Using Evoked Response Potentials to Diagnose Unipolar Major Depression and Bipolar I Depression and Assess Response to Treatment
Brief Title: Brain Network Activation Analysis to Diagnose/Assess Treatment of Unipolar Major Depression and Bipolar I Depression
Acronym: BNA-Mood
Status: Terminated | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, John Zajecka, Associate Professor of Psychiatry, Rush University Medical Center
Other Study IDs: 11122902
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are conducting this study to test the usefulness of a new type of analysis of electroencephalographic (EEG) recordings called brain network activation or BNA. BNA allows to identify patterns of activation in brain networks and to track their changes over time. The investigators want to examine the possible role of brain network activation (BNA) in the diagnosis of mood disorders and predicting improvement over time. The procedure conducted with patients diagnosed with a mood disorder will be compared to people who do not have a mood disorder.

DETAILED DESCRIPTION:
Novel approach to ascertain use of BNA strategy and technology for the use in confirming diagnosis and predicting effect of specific treatment(s)in the various stages of affective/mood disorders. The goal is to develop non-invasive technology to confirm diagnosis via biological outcomes, and to study the preliminary data of predicting response/non-response to specific interventions before clinical effects are shown.

ELIGIBILITY:
Only subjects participating in another specific clinical trial will be invited to participate in this study.

The inclusion/exclusion criteria for this observational study are based on the individual inclusion/exclusion criteria for each of the studies and can be found for each of the studies on this website.

The specific studies and their numbers are found on their individual ClinicalTrials.gov site.

INCLUSION CRITERIA:

Bipolar I, depressed Major depression Meeting all criteria to sign the informed consent for each study included in this study who currently have a major depression (unipolar or bipolarI)

EXCLUSION CRITERIA:

Medically unstable (based on opinion of sponsor and PI Unable to meet the criteria to conform to the Rush University informed consent process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will only enroll subjects who are participating in another specified clinical trial.The inclusion/exclusion criteria will depend on the criteria for each of the studies utilizing subjects with depression or bipolar type I disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2015-08-21 (Actual)

PRIMARY OUTCOMES:
Correlation of changes in BNA with changes in mood symptoms | Beginning of study to end of study
  This is an observational study, so no other outcomes are measured

CONTACTS AND LOCATIONS:
Overall Officials: John M Zajecka, MD, Principal Investigator — RushUMC ; Rush University Medical center